CLINICAL TRIAL: NCT02504489
Title: Randomized Blinded Phase III Assessment of Second or Third-Line Chemotherapy With Docetaxel + Plinabulin Compared to Docetaxel + Placebo in Patients With Advanced Non-Small Cell Lung Cancer and With at Least One Measurable Lung Lesion
Brief Title: Docetaxel + Plinabulin Compared to Docetaxel + Placebo in Patients With Advanced NSCLC
Acronym: DUBLIN-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPI-2358-103
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; NPI 2358; Fumigant 93

STUDY DESIGN:
Who Masked: Participant
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel (D) (Active Comparator): A treatment cycle is 21 days. Treatment will be repeated until disease progression is detected by imaging studies or unacceptable toxicities are encountered. On Day 1, all patients will receive docetaxel 75 mg/m2 by intravenous (IV) infusion over 1 hour. Oral dexamethasone (16 mg, given as 8 mg twice daily) will be given on the day prior to, the day of (Day 1), and the day following docetaxel infusion (Day 2). Antiemetic prophylaxis will be administered according to institutional guideline for docetaxel. Institutional guideline/practice should be followed in the event of infusion/hypersensitivity reaction. Diphenhydramine and dexamethasone infusion may be administered in the event of infusion reaction.
  Interventions: Drug: Docetaxel (D)
- Docetaxel + Plinabulin (DP) (Experimental): The treatment regimen for Docetaxel (D) will be followed for this arm. In addition, on Days 1 and 8 of the 21 day cycle, patients will receive Plinabulin (P) administered via IV infusion over 60 minutes. On Day 1, the infusion begins 2 hours from the starting time of docetaxel infusion, i.e, approximately 60 minutes from the end of docetaxel infusion. On Day 8, patients must be given an anti-emetic prophylactically before the plinabulin infusion. If emesis persists after Day 8, with a grade >1, plinabulin will be reduced to 20 mg/m2. Patients from the DP Arm who stop treatment with docetaxel due to toxicity or another medically acceptable reason, may continue treatment with plinabulin alone as previously described.
  Interventions: Drug: Docetaxel + Plinabulin (DP); Drug: Docetaxel (D)

INTERVENTIONS:
Drug: Docetaxel + Plinabulin (DP) — Docetaxel 75 mg/m2 IV + Plinabulin 30 mg/m2
  Other Names: BPI-2358, NPI-2358
  Arms: Docetaxel + Plinabulin (DP)
Drug: Docetaxel (D) — Docetaxel 75 mg/m2 IV
  Other Names: Taxotere

SUMMARY:
To compare the overall survival of NSCLC patients receiving 2nd- or 3rd-line systemic therapy with docetaxel + plinabulin (DP Arm) to patients treated with docetaxel + placebo (D5W) (D Arm) for advanced or metastatic disease.

Secondary purposes of the study are:

* To compare overall response rate (ORR) of NSCLC patients receiving 2nd- or 3rd-line systemic therapy with docetaxel + plinabulin (DP Arm) to patients treated with docetaxel + placebo (D5W) (D Arm) for advanced or metastatic disease.
* To compare progression free survival (PFS) of NSCLC patients receiving 2nd- or 3rd-line systemic therapy with docetaxel + plinabulin (DP Arm) to patients treated with docetaxel + placebo (D5W) (D Arm) for advanced or metastatic disease.
* To compare incidence of Grade 4 neutropenia (absolute neutrophil count [ANC] < 0.5 × 109/L) on Day 8 (+/- 1 day) of Cycle 1 of NSCLC patients receiving 2nd- or 3rd-line systemic therapy with docetaxel + plinabulin (DP Arm) to patients treated with docetaxel + placebo (D5W) (D Arm) for advanced or metastatic disease.
* To compare 24-month and 36-month OS rate of NSCLC patients receiving 2nd- or 3rd-line systemic therapy with docetaxel + plinabulin (DP Arm) to patients treated with docetaxel + placebo (D5W) (D Arm) for advanced or metastatic disease.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related mortality worldwide. According to the World Health Organization's Global Cancer Observatory, there were an estimated 2.09 million new cases and 1.76 million deaths worldwide in 2018 (GLOBOCAN, 2018, Fact Sheet N⁰39). The lung cancer incidence and mortality in China is relatively high compared to most countries with an estimated 774,323 new cases and 690,567 deaths in 2018 (GLOBOCAN, 2018, Fact Sheet N⁰160 China). In the US, as per the estimates of the National Cancer Institute, there would be about 228,820 new cases and 135,720 deaths from lung cancer in 2020 accounting for approximately 22.4% of all cancer deaths (SEER program, 2020). About 84% of lung cancers are NSCLCs in the US (American Cancer Society, 2020).

The prognosis for patients with advanced or metastatic NSCLC, either at initial diagnosis or recurrence, remains grim. The standard of care has been chemotherapy with agents including platinum analogs, taxanes, vinca alkaloids, and pemetrexed with vascular endothelial growth factor inhibitors and for patients with appropriate disease genotypes, epidermal growth factor receptor (EGFR) inhibitors or anaplastic lymphoma kinase (ALK) inhibitors.

First-line Therapy: For patients without specific molecular target, first-line therapy is usually a programmed cell death protein 1 (PD-1)-inhibitor or a platinum-containing, double agent regimen. Platinum can be either cisplatin or carboplatin, and the most commonly used drugs combined with platinum include paclitaxel, docetaxel, gemcitabine, and vinorelbine; other drugs such as irinotecan, etoposide, and vinblastine.

The arrival of immunotherapy with the PD-1 inhibitor pembrolizumab effectively changed the first-line standard. Pembrolizumab is very effective, with a long Duration of Response (DoR), however response rates remain suboptimal (approximately 45% in first line [Keytruda® Prescribing Information. 2020]). Most patients will eventually fail first line therapy and docetaxel remains a valid treatment option when NSCLC patients fail to respond to targeted or immune-based therapies or become refractory to such therapies.

For patients intolerant to platinum-containing regimens, platinum-free double-agent chemotherapy regimens are used as an alternative. For patients with an Eastern Cooperative Oncology Group score of 2 and elderly patients, single-agent or double agent regimens are recommended. Approval has been obtained in China for the single agent gefitinib to be used in first-line treatment of locally advanced or metastatic NSCLC patients with sensitive mutation of EGFR tyrosine kinase gene.

Second-line Therapy: Drugs used for second-line treatment include docetaxel, pemetrexed, EGFR-tyrosine kinase inhibitor (TKI) for EGFR mutant patients, and the checkpoint inhibitors (such as nivolumab and pembrolizumab).

Several second-line treatment drugs and regimens (docetaxel, pemetrexed, and ramucirumab combined with docetaxel) have been approved as single agents or combination for second-line therapy for locally advanced or metastatic NSCLC with EGFR wild type with limited efficacy, characterized by limited clinical improvement or overall survival (OS). EGFR wild type represents around 85% of western NSCLC population, and around 70% of Asian NSCLC population. Checkpoint inhibition with PD 1/programmed death-ligand 1 (PD-L1) inhibitors in combination with chemotherapy or other checkpoint inhibitors have moved into first line and are increasingly not an option for 2nd/3rd line. This has created a situation where docetaxel-based regimens have become standard-of-care in 2nd/3rd line NSCLC. Therefore, the evaluation of plinabulin combined with docetaxel versus docetaxel alone has become highly relevant.

Docetaxel, a taxane, binds to and stabilizes tubulin, thereby inhibiting microtubule disassembly resulting in cell cycle arrest at the G2/M phase and subsequent cell death. In patients with NSCLC, previously treated with a platinum-based chemotherapy, second-line therapy with docetaxel afforded a median OS in the range from 5.7 to 7.5 months (Fossella, 2000; Shepherd, 2000). The most common AEs included infections, neutropenia, anemia, febrile neutropenia (FN), hypersensitivity, thrombocytopenia, neuropathy, dysgeusia, dyspnea, constipation, anorexia, nail disorders, fluid retention, asthenia, pain, nausea, diarrhea, vomiting, mucositis, alopecia, skin reactions, and myalgia (Taxotere Prescribing Information, 2020). Since the approval of docetaxel in 1999 as the second-line treatment for advanced or metastatic NSCLC, other drugs, namely pemetrexed and erlotinib, have been approved for the same indication. However, despite the availability of newer treatments, patient survival has not improved over that achieved with docetaxel. The OS in these studies was found to remain in the range of 5.6 to 8.3 months (Hanna et al., 2004; Kim et al., 2008; Shepherd et al., 2005).

A retrospective analysis of the plinabulin Phase 2 study suggests that plinabulin prolongs survival in NSCLC patients with measurable lung tumors. The expectation is that patients with a measurable lung lesion may still harbor antigens that are immunogenic, thus capable of still stimulating the immune system. Docetaxel treatment is expected to release these immunogens and plinabulin is expected to enhance presentation of these immunogens via dendritic cell activation, to the T-cell repertoire.

This plinabulin study investigates the efficacy and safety of plinabulin and docetaxel combination in patients with EGFR wild type NSCLC and progressing tumors requiring second- or third- line therapy for advanced or metastatic disease after failing a platinum-containing regimen. The primary endpoint is OS, with docetaxel monotherapy as an active comparator.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Males and females ≥ 18 years of age
2. ECOG performance status ≤ 2.
3. Histopathologically or cytologically confirmed non-squamous or squamous NSCLC.
4. Disease progression during or after treatment with one or two treatment regimen(s) Treatment regimens can be chemotherapy, targeted therapy, biological therapy, or immunotherapy for advanced (Stage IIIB) or metastatic disease (Stage IV). Modification of a regimen to manage toxicity with a different drug does not constitute a new regimen. Maintenance therapy following platinum-based chemotherapy is not considered as a separate regimen. Adjuvant or neoadjuvant chemotherapy and/or chemo-radiation for early stage disease do not count as prior systemic therapy. Prior radiation therapy is not exclusionary. Prior immunotherapy with a PD-1/PD-L1 inhibitor is not exclusionary. Prior treatment for advanced or metastatic disease must have included a platinum-based regimen. (Treatment of early stage disease [Stage IIIA or earlier] with a platinum-containing therapy does not count).
5. Patients with active brain metastasis or leptomeningeal involvement with brain metastases who are asymptomatic, and whose lesions by imaging are at least stable and without interim development of new lesions for at least 4 weeks may be enrolled. Patients who require continued therapy with steroid medication for management for their brain metastases are eligible; dosing must be stable for at least 4 weeks prior to randomization;
6. Patients must have at least one measurable lung lesion of ≥10 mm by CT or MRI per RECIST 1.1 criteria. Radiographic tumor assessment is to be performed within 28 days prior to randomization;
7. All patients with non-squamous NSCLC must have been tested for 19 deletion and exon 21 L858R substitution mutation. Only patients without EGFR sensitizing mutations are eligible, and they must have progressed on platinum-based chemotherapy. Patients with known ALK-rearrangements should be treated with an appropriate tyrosine kinase inhibitor (TKI) before entering the study. The TKI regimen would count as a line of treatment.
8. All adverse events of any prior systemic therapy, surgery, or radiotherapy, must have resolved to CTCAE (v4.03) Grade ≤2, except for neurological adverse events that must have resolved to Grade ≤1;
9. The following laboratory results from the central laboratory within 14 days prior to Cycle 1 Day 1 study drug administration.

   * Hemoglobin ≥9 g/dL independent of transfusion or growth factor support;
   * Absolute neutrophil count ≥1.5 x 109/L independent of growth factor support;
   * Platelet count ≥100 x 109/L independent of transfusion or growth factor support;
   * Serum total bilirubin ≤ ULN, unless the patient has a diagnosis of Gilbert's disease in which case serum bilirubin ≤3.0 times ULN;
   * AST and ALT ≤2.5 x ULN (≤1.5 x ULN if alkaline phosphatase is >2.5 x ULN);
   * Serum creatinine ≤1.5 x ULN;
10. Life expectancy more than 12 weeks;
11. Female patients of childbearing potential have a negative pregnancy test at baseline. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

    1. Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.
    2. Sexually active women of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.
    3. For male patients who are sexually active and who are partners of premenopausal women: agreement to use two forms of contraception as in criterion 11b above during the treatment period and for at least 3 months after the last dose of study drug.
12. Signed informed consent.

EXCLUSION CRITERIA: Patients with any of the following:

1. Administration of chemotherapy, immunotherapy, biological, targeted, or radiation therapy or investigational agent (therapeutic or diagnostic) within 3 weeks prior to receipt of study medication. Major surgery, other than diagnostic surgery, within 4 weeks before first study drug administration.
2. Significant cardiac history:

   * History of myocardial infarction or ischemic heart disease within 1 year (within a window of 18 days) before first study drug administration;
   * Uncontrolled arrhythmia;
   * History of congenital QT prolongation;
   * ECG findings consistent with active ischemic heart disease;
   * New York Heart Association Class III or IV cardiac disease;
   * Uncontrolled hypertension: blood pressure consistently greater than 150 mm Hg systolic and 100 mm Hg diastolic in spite of antihypertensive medication.
3. Patients who have received prior treatment with docetaxel.
4. Prior transient ischemic attack or cerebrovascular accident within the past year (within an 18-day window). Any neurologic toxicities ≥ Grade 2 within 3 weeks of randomization.
5. History of hemorrhagic diarrhea, inflammatory bowel disease or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
6. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
7. Known infection with human immunodeficiency virus (HIV) or active hepatitis A, B, or C.
8. Known prior hypersensitivity reaction to any product containing polysorbate 80, polyoxyethylene 15 hydroxystearate/Macrogol 15 hydroxystearate (Solutol HS 15/ Kolliphor HS 15).
9. Female subject who is pregnant or lactating.
10. Second malignancy unless in remission for >5 years. (Non-melanoma skin cancer or carcinoma in situ of the cervix treated with curative intent is not exclusionary).
11. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include uncontrolled diabetes, infection requiring parenteral anti-infective treatment, liver failure, any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent form.
12. Unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-05-23 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Mid-February 2021 (Approximately 2 years after study initiation)
  Overall survival of NSCLC patients receiving 2nd- or 3rd-line systemic therapy

SECONDARY OUTCOMES:
ORR | Approximately 2 years after study initiation.
  Overall response rate
PFS | Approximately 2 years after study initiation.
  Progress-free survival
Severe Neutropenia | Day 8 of Cycle 1
  Percent of patients without severe neutropenia on Day 8 of Cycle 1
Month 24 OS Rate | 24-month after study initiation
  To compare 24-month overall survival rate
Month 36 OS Rate | 36 month after study initiation
  To compare 36-month overall survival rate
DoR | Approximately 2 years after study initiation.
  Duration of response
Quality of Life (EORTC QLQ-C30) | Approximately 2 years after study initiation.
  Average Quality of Life score over all observed weeks (scale 0 - 30, higher value represents better outcome)
Q-TWiST | Approximately 2 years after study initiation.
  To compare the mean difference in quality-adjusted time without symptoms of disease and toxicity
QoL (QLQ-LC13) | Approximately 2 years after study initiation.
  To compare the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 global health status/QoL and the combined symptom scales/items (excluding financial difficulties)
Proportion of patients who received docetaxel | During 1st 21-day cycle
  To compare proportion of patients who received docetaxel >8 cycles, >10 cycles, and >12 cycles
Month 18 OS Rate | 18 month after study initiation
  To compare 18-month overall survival rate
RDI | First 4, 6, 8, 10, and 12 cycles
  To compare relative dose intensity [where dose intensity is defined as dose in mg/m2/week] of docetaxel
Month 12 OS Rate | 12 month after study initiation
  To compare 12-month overall survival rate

CONTACTS AND LOCATIONS:
Locations (57):
- United States (19):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Innovative Clinical Research Institute, Whittier, California
  - Memorial Health Care System, Colorado Springs, Colorado
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Peachtree Hematoloy-Oncology Consultants, PC, Atlanta, Georgia
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Kansas University Medical Center, Westwood, Kansas
  - University of Louisville-Brown Cancer Center, Louisville, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Central Care Cancer Center, Bolivar, Missouri
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Toledo Cancer Center, Toledo, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Cookeville Regional Medical Center Cancer Center, Cookeville, Tennessee
- Australia (9):
  - Blacktown Cancer Centre, Blacktown, New South Wales
  - Border Medical Oncology Research Unit, East Albury, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Adult Mater Hospital, South Brisbane, Queensland
  - Peninsula and South East Oncology, Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Perth Oncology/Mount Hospital, Perth, Western Australia
  - St John of God Hospital, Subiaco, Subiaco, Western Australia
- China (29):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guizhou Provincial Hospital, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical Unive, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South Unive, Changsha, Hunan
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Jiangxi Provincial Tumor Hospital, Nanchang, Jiangxi
  - Jilin Province Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong U, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shangdong
  - 527-Linyi Cancer Hospital, Linyi, Shangdong
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Shanghai Chest Hospital, Shanghai Jiaotong Univers, Shanghai, Shanghai Municipality
  - The Fifth People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical Univ, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han B, Feinstein T, Shi Y, Chen G, Yao Y, Hu C, Shi J, Feng J, Wu H, Cheng Y, Guo QS, Jie Z, Ye F, Zhang Y, Liu Z, Mao W, Zhang L, Lu J, Zhao J, Bazhenova L, Ruiz J, Kloecker GH, Sujith KR, Oliff IA, Wong M, Liu B, Wu Y, Huang L, Sun Y; DUBLIN-3 study group. Plinabulin plus docetaxel versus docetaxel in patients with non-small-cell lung cancer after disease progression on platinum-based regimen (DUBLIN-3): a phase 3, international, multicentre, single-blind, parallel group, randomised controlled trial. Lancet Respir Med. 2024 Oct;12(10):775-786. doi: 10.1016/S2213-2600(24)00178-4. Epub 2024 Sep 9. PMID 39265599
- See also: BeyondSpring Pharmaceuticals, Inc. Web-site — http://beyondspringpharma.com